CLINICAL TRIAL: NCT02988518
Title: Evaluation of a Cognitive Remediation Program on Patients With Bipolar Disorders, With Memory Complaints
Brief Title: Cognitive Remediation on Patients With Bipolar Disorder and Memory Complaints
Acronym: COGMED
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UF 9418; 2014-A00825-42 (Other: Agence nationale de Sécurité des Médicaments)
Record Dates: First submitted 2016-08-01; First posted 2016-12-09 (Estimated); Last update posted 2016-12-09 (Estimated); Status verified 2016-07

CONDITIONS: Patient With Bipolar Disorder; Euthymic Status; Wirh Memory Complaints
Keywords: Psychiatry; Bipolar disorder; Memory complaints; Global functioning; Cognitive remediation; Working memory
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- COGMED program (Experimental): Cognitive remediation using COGMED program on bipolar euthymic patients with memory complaints
  Interventions: Behavioral: COGMED program

INTERVENTIONS:
Behavioral: COGMED program — Patient should connect on his computer at home, 5 times a week, for 5 weeks. Every day, the patient has to do 8 exercises for a total duration of 30 to 45 minutes.
  In total, the patient will have to complete 25 sessions. The difficulty level of the proposed items adjust automatically to the patient's maximum capacity to compel him to provide a cognitive effort. A progression index assesses the progress made by the patient.
  Every week, the investigator will call the patient for 10 minutes in order to gather the patient's feelings, his difficulties, provide some advice and encourage him.
  The investigator will have to analyze the results of curves available for each event, as well as the patient's progress index.

SUMMARY:
Bipolar disorder is a major health concern. Intercritical periods are marked with residual symptoms, both thymic and cognitive, which affects quality of life of patients, but also the quality of observance. The implementation of cognitive remediation programs could be interesting. The aim of this study is to evaluate the overall performance on euthymic bipolar patients with memory complaints included in the program named "COGMED", targeting the working memory.

The impact of this program on compliance, quality of life, and memory complaints will be evaluated.

The investigator will measure whether there is a correlation between working memory and overall performances.

Finally, the investigator will try to achieve a profile of bipolar patients in whom the Cogmed program is particularly effective on a plan of overall performance.

DETAILED DESCRIPTION:
Patients with bipolar disorder and memory complaints will be recruited.

Two visits :

1. at baseline (V0) : the investigator evaluate bipolar disorder, treatment, mood, quality of life, global functioning, and memory complaints. Patients also have a neuropsychological assessment. The COGMED program is proposed to patients with memory complaints and explain by the investigator
2. 4-6 weeks after the end of the program (11-13 weeks after V1) : the same evaluation is realized to compare score before and after the program of cognitive remediation.

Between the two visits the patient will benefit of COGMED program, at home, during 5 weeks.

COGMED is a remediation cognitive program, based on working memory, consisting on daily exercises at home on a computer.

ELIGIBILITY:
Inclusion criteria:

* Being diagnosed bipolar according to the Diagnostic and Statistical Manual of Mental Disorders - IV (DSM-IV) criteria
* Memory complaints or overall performance alterations according to the memory scale (MEM III Wechsler memory scale - third edition)
* Being euthymic at the inclusion according to Montgomery-Asberg Depression Rating Scale (MADRS < 12) and Young Mania Rating Scale (YMRS < 6)
* Not being treated with electroconvulsive therapy for the last year
* Not having drug-dependance or drug-abuse for the last six months
* Having a computer with internet and a cellphone at home
* Having signed informed consent
* Able to understand nature, aims and methodology of the study

Exclusion criteria:

* Patient on protective measures (guardianship or trusteeship)
* Deprived of liberty subject (judicial or administrative decision)

Ages: 18 Months to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2014-07; Primary Completion 2017-11 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Evolution of the global functioning between the inclusion and the end of the program | At 4 weeks
  evaluation of variation of global functioning will be realized by the Functioning Assessment Short Test (FAST) scale after COGMED program.
Evolution of the global functioning between the inclusion and the end of the program | At 6 weeks
  evaluation of variation of global functioning will be realized by the Functioning Assessment Short Test (FAST) scale after COGMED program

SECONDARY OUTCOMES:
Observance | At the inclusion and 4 to 6 weeks until the end of the program COGMED (11 to 13 weeks after inclusion)
  Evaluation of variation of patient's compliance by Medication Adherence Rating Scale (MARS) score after COGMED program.
Quality of life | At the inclusion and 4 to 6 weeks until the end of the program COGMED (11 to 13 weeks after inclusion)
  Evaluation of variation of quality of life by Short Form (36) Health Survey (SF-36) score after COGMED program.
Correlation between working memory and global functioning | At the inclusion and 4 to 6 weeks until the end of the program COGMED (11 to 13 weeks after inclusion)
  Searching a statistical correlation between global functioning (using FAST) and working memory (using neuropsychological tests)
Memory complaints | At the inclusion and 4 to 6 weeks until the end of the program COGMED (11 to 13 weeks after inclusion)
  Variations on memory complaints will be evaluated by Mac Nair Scale score before and after COGMED program.

CONTACTS AND LOCATIONS:
Locations (1):
- Montpellier University Hospital, Montpellier, France

IPD SHARING:
Plan to Share IPD: No